CLINICAL TRIAL: NCT02832843
Title: Elucidation of Genetic Susceptibility of Patients With Nontuberculous Mycobacterial Lung Disease Using Genome-Wide Association Study
Brief Title: Genome-Wide Association Study in Patients With Nontuberculous Mycobacterial Lung Disease
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: H-1605-111-763
Record Dates: First submitted 2016-07-03; First posted 2016-07-14 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Extraction of DNA will be conducted from serum of patients with NTM lung disease. For controls, preexisting dataset of GWAS will be used.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NTM lung disease: Patients with NTM lung disease satisfying American Thoracic Society guidelines
- Healthy control: The age-, sex-matched control subjects without pulmonary diseases

SUMMARY:
The aim of this study was to elucidate genetic susceptibility of patients with nontuberculous mycobacterial lung disease using genome-wide association study.

DETAILED DESCRIPTION:
Nontuberculous mycobacteria (NTM) are ubiquitous environmental organisms. NTM lung disease is increasing, however, genetic susceptibility of patients with the disease have not been identified. To elucidate the genetic susceptibility of NTM lung disease, the investigators perform a genome-wide association study (GWAS) including patients with NTM lung disease and healthy controls (case : control = 1 : 3). The age-, sex-matched control group will be recruited from the Korean Healthy Twin Study.

ELIGIBILITY:
Inclusion Criteria:

* Case: Patients with NTM lung disease satisfying diagnostic criteria suggested by American Thoracic Society
* Control: Healthy subjects enrolled in the Korean Healthy Twin Study

Exclusion Criteria:

* Case: none
* Control: 1) Subjects who have respiratory symptoms including cough and sputum 2) Subjects who have abnormalities on chest radiography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with NTM lung diseases and healthy control
Sampling Method: Non-Probability Sample
Enrollment: 2808 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Finding of single nucleotide polymorphisms (SNPs) associated with the risk of NTM lung disease compared with controls | Baseline
  To identify SNPs related to NTM lung disease using logistic regression after controlling for confounders (GWAS statistical significance threshold, P < 5.00*E-08)

SECONDARY OUTCOMES:
Finding of SNPs associated with the risk of severe NTM lung disease compared with controls | Baseline
  To identify SNPs related to severe NTM lung disease compared with controls using logistic regression after controlling for confounders (GWAS statistical significance threshold, P < 5.00*E-08)
Finding of SNPs associated with the risk of severe NTM lung disease compared with mild NTM lung disease | Baseline
  To identify SNPs related to severe NTM lung disease compared with mild NTM lung disease using logistic regression after controlling for confounders (GWAS statistical significance threshold, P < 5.00*E-08)
Finding of SNPs associated with the risk of Mycobacterium avium complex lung disease versus M. abscessus lung disease versus controls | Baseline
  To identify SNPs related to Mycobacterium avium complex lung disease versus M. abscessus lung disease versus controls using multinomial logistic regression after controlling for confounders (GWAS statistical significance threshold, P < 5.00*E-08)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park YS, Lee CH, Lee SM, Yang SC, Yoo CG, Kim YW, Han SK, Shim YS, Yim JJ. Rapid increase of non-tuberculous mycobacterial lung diseases at a tertiary referral hospital in South Korea. Int J Tuberc Lung Dis. 2010 Aug;14(8):1069-71. PMID 20626955
- [Background] Yim JJ, Kim HJ, Kwon OJ, Koh WJ. Association between microsatellite polymorphisms in intron II of the human Toll-like receptor 2 gene and nontuberculous mycobacterial lung disease in a Korean population. Hum Immunol. 2008 Sep;69(9):572-6. doi: 10.1016/j.humimm.2008.06.003. Epub 2008 Jul 3. PMID 18602432
- [Background] Kim RD, Greenberg DE, Ehrmantraut ME, Guide SV, Ding L, Shea Y, Brown MR, Chernick M, Steagall WK, Glasgow CG, Lin J, Jolley C, Sorbara L, Raffeld M, Hill S, Avila N, Sachdev V, Barnhart LA, Anderson VL, Claypool R, Hilligoss DM, Garofalo M, Fitzgerald A, Anaya-O'Brien S, Darnell D, DeCastro R, Menning HM, Ricklefs SM, Porcella SF, Olivier KN, Moss J, Holland SM. Pulmonary nontuberculous mycobacterial disease: prospective study of a distinct preexisting syndrome. Am J Respir Crit Care Med. 2008 Nov 15;178(10):1066-74. doi: 10.1164/rccm.200805-686OC. Epub 2008 Aug 14. PMID 18703788
- [Background] Lee AR, Lee J, Choi SM, Seong MW, Kim SA, Kim M, Chae KO, Lee JS, Yim JJ. Phenotypic, immunologic, and clinical characteristics of patients with nontuberculous mycobacterial lung disease in Korea. BMC Infect Dis. 2013 Nov 25;13:558. doi: 10.1186/1471-2334-13-558. PMID 24274658
- [Background] Kim J, Seong MW, Kim EC, Han SK, Yim JJ. Frequency and clinical implications of the isolation of rare nontuberculous mycobacteria. BMC Infect Dis. 2015 Jan 9;15:9. doi: 10.1186/s12879-014-0741-7. PMID 25572753
- [Background] Kwak N, Lee CH, Lee HJ, Kang YA, Lee JH, Han SK, Yim JJ. Non-tuberculous mycobacterial lung disease: diagnosis based on computed tomography of the chest. Eur Radiol. 2016 Dec;26(12):4449-4456. doi: 10.1007/s00330-016-4286-6. Epub 2016 Mar 5. PMID 26945763
- [Background] Hill AV. Evolution, revolution and heresy in the genetics of infectious disease susceptibility. Philos Trans R Soc Lond B Biol Sci. 2012 Mar 19;367(1590):840-9. doi: 10.1098/rstb.2011.0275. PMID 22312051
- [Background] Sung J, Cho SI, Lee K, Ha M, Choi EY, Choi JS, Kim H, Kim J, Hong KS, Kim Y, Yoo KY, Park C, Song YM. Healthy Twin: a twin-family study of Korea--protocols and current status. Twin Res Hum Genet. 2006 Dec;9(6):844-8. doi: 10.1375/183242706779462822. PMID 17254419
- [Background] Li Y, Willer CJ, Ding J, Scheet P, Abecasis GR. MaCH: using sequence and genotype data to estimate haplotypes and unobserved genotypes. Genet Epidemiol. 2010 Dec;34(8):816-34. doi: 10.1002/gepi.20533. PMID 21058334
- [Background] Howie BN, Donnelly P, Marchini J. A flexible and accurate genotype imputation method for the next generation of genome-wide association studies. PLoS Genet. 2009 Jun;5(6):e1000529. doi: 10.1371/journal.pgen.1000529. Epub 2009 Jun 19. PMID 19543373
- [Background] 1000 Genomes Project Consortium; Abecasis GR, Altshuler D, Auton A, Brooks LD, Durbin RM, Gibbs RA, Hurles ME, McVean GA. A map of human genome variation from population-scale sequencing. Nature. 2010 Oct 28;467(7319):1061-73. doi: 10.1038/nature09534. PMID 20981092
- [Background] Ritchie MD, Hahn LW, Roodi N, Bailey LR, Dupont WD, Parl FF, Moore JH. Multifactor-dimensionality reduction reveals high-order interactions among estrogen-metabolism genes in sporadic breast cancer. Am J Hum Genet. 2001 Jul;69(1):138-47. doi: 10.1086/321276. Epub 2001 Jun 11. PMID 11404819